CLINICAL TRIAL: NCT04279041
Title: In-vitro and In-vivo Comparative Evaluation of Rotary Fanta and Zunba Files in Root Canal Preparation of Infected Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmad Elheeny (Other)
Responsible Party: Sponsor-Investigator, Ahmad Elheeny, clinical professor, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 260
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Root Canal Preparation of Infected Primary Molars
MeSH Terms: interventions — Root Canal Preparation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fanta and Zunba rotatory files (Experimental): Fanta and Zunba rotatory files
  Interventions: Procedure: root canal preparation
- manual K-files (Active Comparator): manual K-files
  Interventions: Procedure: root canal preparation

INTERVENTIONS:
Procedure: root canal preparation — root canal preparation

SUMMARY:
Adequate shaping and cleaning, followed by a good coronal seal, are prerequisites for a favorable outcome. The goal of root canal preparation is to create optimized canal geometry to allow effective irrigation and obturation with preservation of the original canal morphology.

The aim of current study is to evaluate the effectiveness of Fanta and Zunba rotatory instruments in cleaning of infected root canal of primary molars to those instrumented with manual K-files.

ELIGIBILITY:
Inclusion Criteria:

* Class I or II according to American Society of Anesthesiologists (ASA)
* Necrotic pulp tissues which may be asymptomatic or manifested with dull ache pain
* Pathological tooth mobility
* Percussion sensitivity
* Swelling close to involved tooth accompanied with or without fistula
* The extension of radiolucency at the furcation area did not exceed half of the space between the furcation and the permanent successor
* No internal root resorption
* External root resorption (Physiologic or pathologic) limited to apical third and with at least two-third root intact

Exclusion Criteria:

* Uncooperativeness of child and/or parents or caregiver's behavior.
* Unrestorable tooth.
* Presence of calcific metamorphosis inside root canals.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
clinical success rate | 12 month
  Presence or abscnce (+/-) of pain, mobility and/or fistulous tract
radiographic success rate | 12 month
  Presence or abscnce (+/-) of periapical rdiolucency

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University, Minya, Egypt

REFERENCES:
- [Derived] Abd El Fatah YAM, Elheeny AAH, Ashraf Abd-Elsabour MA, Ali Khattab NM. Clinical and radiographic outcomes of pulpectomy in primary teeth using two rotary file systems compared with manual files: a cost-effectiveness analysis. BMC Oral Health. 2025 Jul 4;25(1):1093. doi: 10.1186/s12903-025-06508-y. PMID 40616048